CLINICAL TRIAL: NCT04792567
Title: An Open-label Multicenter Study to Assess Response to SARS-CoV-2 modRNA Vaccines in Participants With Secondary Progressive Multiple Sclerosis Treated With Mayzent (Siponimod)
Brief Title: Exploring the Immune Response to SARS-CoV-2 modRNA Vaccines in Patients With Secondary Progressive Multiple Sclerosis (AMA-VACC)
Acronym: AMA-VACC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBAF312ADE03; 2020-005752-38 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: COVID-19; SARS-CoV-2 mRNA vaccine; Siponimod; Secondary Progressive Multiple Sclerosis; SPMS; adult; MS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; COVID-19 | interventions — siponimod; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Siponimod - continuous (Experimental): Continuous treatment with siponimod (oral, daily, dose depending on CYP2C9 genotype: 2mg or 1 mg) during SARS-CoV-2 mRNA vaccination
  Interventions: Drug: BAF312; Biological: BNT162; Biological: mRNA-1273
- Siponimod- interrupted (Experimental): Siponimod (oral, daily, dose depending on CYP2C9 genotype: 2mg or 1 mg) with treatment interruption (for approx. 2-3 months) for the purpose of a SARS-CoV-2 mRNA vaccination
  Interventions: Drug: BAF312; Biological: BNT162; Biological: mRNA-1273
- Comparator (Active Comparator): Baseline DMTs or no treatment during SARS-CoV-2 mRNA vaccination
  Interventions: Drug: Baseline disease modifying therapies (DMTs); Biological: BNT162; Biological: mRNA-1273

INTERVENTIONS:
Drug: BAF312 — taken orally once per day (dose depends on CYP2C9 genotype)
  Other Names: Siponimod
  Arms: Siponimod - continuous; Siponimod- interrupted
Drug: Baseline disease modifying therapies (DMTs) — DMTs: Dimethylfumarate, glatirameracetate, interferon, teriflunomode according to respective SmPC
  Arms: Comparator
Biological: BNT162 — Administerd according to the respective EU SmPC at the discretion of the treating physician independent of AMA-VACC. If suggested by local regulations and performed as part of clinical routine any type of booster/refresher vaccination (e.g. mRNA, vector, peptide) was allowed in this study.
  Other Names: Comirnaty®
Biological: mRNA-1273 — Administerd according to the respective EU SmPC at the discretion of the treating physician independent of AMA-VACC. If suggested by local regulations and performed as part of clinical routine any type of booster/refresher vaccination (e.g. mRNA, vector, peptide) was allowed in this study
  Other Names: Spikevax®

SUMMARY:
The purpose of this study was to understand whether participants could mount an immune response to SARS-CoV-2 modRNA vaccines administered either during continuous siponimod treatment or during a treatment break versus while on treatment with first-line DMTS or no current MS treatment..

DETAILED DESCRIPTION:
This was a three cohort, multicenter, open-label, study of 60 planned (optionally up to 90) multiple sclerosis (MS) patients who were on treatment with siponimod or a first-line disease modifying therapy (DMT) or without MS treatment planning to undergo a SARS-CoV-2 modRNA vaccination as part of clinical routine.

* The first cohort enrolled participants who did not interrupt their siponimod therapy for the purpose of a SARS-CoV-2 modRNA vaccination.
* The second cohort enrolled participants who interrupted their siponimod therapy for the purpose of a SARS-CoV-2 modRNA vaccination for approximately 2-3 months
* The third cohort enrollled participants who received modRNA vaccination while on treatment with the following first-line DMTs (dimethylfumarate, glatirameracetate, interferons, teriflunomide) or no current treatment in clinical routine.

The study consists of a screening period, vaccination period and investigational period. During the screening period of up to one month eligibility and SARS-CoV-2 antibodies at baseline were assessed. The 3-4 week vaccination period started with first dose of modRNA vaccine on Day 1 and ended with second dose of modRNA vaccine 3-4 weeks after first dose depending on EU SmPC.

The investigational period lasted 12 months, during which blood samples for primary and secondary endpoint analyses were drawn at 1 week (Visit 1), 1 Month (Visit 2) and 6 months (Visit 3) after completion of vaccination (i.e. second dose of vaccine). 12 months after completion of vaccination a COVID-19 follow-up call was scheduled.

As patients were treated according to clinical routine, the start of treatment was defined as the date the informed consent was signed.

Booster vaccinations were allowed as per local regulations, physician's discretion and as part of clinical routine. This booster may have been any type of SARS-CoV2 vaccine and introduction of a treatment break for the purpose of booster vaccination was at the discretion of the treating physician or patient for all three cohorts. In case of booster vaccinations an additional blood sample was collected 1 month after the booster vaccination (booster Visit).

The planned study duration for each participant was 56-64 weeks, depending on the length of the screening period.

The study investigated the development of functional anti-SARS-CoV-2 antibodies and T-cell titers for six months after the participants' vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Secondary Progressive Multiple Sclerosis (SPMS) diagnosis or with Relapsing Remitting Multiple Sclerosis (RRMS) at risk to develop SPMS (at the discretion of the treating physician)
* on stable MS treatment (Siponimod, dimethylfumarate, glatirameracetate, interferon, teriflunomode) or no current treatment
* no recent treatment changes

Exclusion Criteria:

* prior or current COVID-19 disease
* SARS-CoV-2 antibodies at screening Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (10):
  - Novartis Investigative Site, Mittweida, Saxony
  - Novartis Investigative Site, Bogen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Ulm

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] Ziemssen T, Groth M, Rauser B, Bopp T. Assessing the immune response to SARS-CoV-2 mRNA vaccines in siponimod-treated patients: a nonrandomized controlled clinical trial (AMA-VACC). Ther Adv Neurol Disord. 2022 Nov 8;15:17562864221135305. doi: 10.1177/17562864221135305. eCollection 2022. PMID 36381503
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1559

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants screened were enrolled, there were no screen failures.
Groups:
- DMT or no MS Treatment: Baseline disease modifying treatments (DMTs) or no multiple sclerosis treatment during SARS-CoV-2 mRNA vaccination
Period: Overall Study
Arm/Group | Siponimod - Continuous | Siponimod- Interrupted | DMT or no MS Treatment
Started | 17 | 4 | 20
Completed | 17 | 4 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Siponimod - Continuous | Siponimod- Interrupted | DMT or no MS Treatment | Total
Number analyzed (Participants) | 17 | 4 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (5.8) | 55.8 (2.2) | 48.6 (12.9) | 51.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16 | 32
  Male | 4 | 1 | 4 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 14 | 3 | 17 | 34
  African | 0 | 0 | 0 | 0
  Other | 1 | 1 | 2 | 4
  Missing | 2 | 0 | 1 | 3
Multiple sclerosis diagnosis [Count of Participants; unit: Participants] — The diagnosis of type of multiple sclerosis at baseline.
  Participants
    SPMS Secondary progressive multiple sclerosis | 14 | 1 | 2 | 17
    RRMS Relapsing remitting multiple sclerosis | 0 | 0 | 11 | 11
    Active SPMS (with acute exacerbation or progression) | 3 | 3 | 0 | 6
    MS Multiple sclerosis, not specified | 0 | 0 | 6 | 6
    Active RRMS (with acute exacerbation or progression) | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroconversion One Week After Receiving Second Vaccine (EAS)
Description: Participants who had detectable SARS-CoV-2 serum functional antibodies one week after second dose of vaccine.
Time Frame: At 1 week after vaccination period (defined as 1 week after second dose of vaccine)
Population: Efficacy analysis set (EAS) - all participants who had a valid primary endpoint (i. e. determination of functional antibodies to SARS-CoV-2 at Week 1 after second dose of vaccine)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Siponimod - Continuous | Siponimod- Interrupted | DMT or no MS Treatment
Number analyzed (Participants) | 17 | 4 | 20
percentage of participants | 52.9 [27.8 to 77.0] | 75.0 [19.4 to 99.4] | 90.0 [68.3 to 98.8]

2. Secondary Outcome: SARS-CoV-2 Functional Antibodies (% Inhibition) by Visits (SAF/EAS)
Description: Measurement of antibody-mediated blockage (i.e. presence of functional SARS-CoV-2 antibodies) was performed to quantify functional SARS-CoV-2 neutralizing antibodies and was calculated as % inhibition to the in-assay control.
Time Frame: Baseline; Week 1, Month 1 and Month 6 after second dose of vaccine; 1 month after booster (up to Month 12 after second dose of vaccine)
Population: Safety analysis set (received any study drug) and efficacy analysis set (participants with a valid primary endpoint)
Measure: Mean (Standard Deviation); unit: antibody titer levels (% inhibition)
Arm/Group | Siponimod - Continuous | Siponimod- Interrupted | DMT or no MS Treatment
Number analyzed (Participants) | 17 | 4 | 20
antibody titer levels (% inhibition)
  Screening n=17,4,20 | -3.8 (5.0) | -0.3 (11.1) | -2.6 (8.2)
  Visit 1/Week 1 n=17,4,20 | 38.1 (34.8) | 64.0 (41.8) | 82.6 (26.7)
  Visit 2/Month 1 n=16,4,20: number analyzed (Participants) | 16 | 4 | 20
  Visit 2/Month 1 n=16,4,20 | 40.1 (27.2) | 87.5 (16.4) | 86.8 (21.5)
  Visit 3/Month 6 n=16,4,20: number analyzed (Participants) | 16 | 4 | 20
  Visit 3/Month 6 n=16,4,20 | 43.2 (32.8) | 68.3 (34.5) | 77.3 (27.1)
  1 Month after booster n=16,4,18: number analyzed (Participants) | 16 | 4 | 18
  1 Month after booster n=16,4,18 | 62.3 (30.3) | 96.5 (2.4) | 96.8 (2.8)

3. Secondary Outcome: Number of Patients Reactive to INFg or IL-2 SARS-CoV-2 by Visit SAF/EAS
Description: The release of IFNg or IL-2 after stimulation with a SARS-CoV-2/PAN corona peptide-mix measured by enzyme-linked immunosorbent spot (ELIspot) assay from peripheral blood mononuclear cells indicates the presence of SARS-CoV-2 reactive T-cells, i.e. a T-cell response.
Time Frame: as for outcome 2
Population: Safety analysis set (received any study drug) and efficacy analysis set (participants with a valid primary endpoint)
Measure: Number; unit: participants
Arm/Group | Siponimod - Continuous | Siponimod- Interrupted | DMT or no MS Treatment
Number analyzed (Participants) | 17 | 4 | 20
participants
  Screening reactive n=17,4,20 | 0 | 0 | 1
  Screening not reactive n=17,4,20 | 10 | 3 | 19
  Screening missing value n=17,4,20 | 7 | 1 | 0
  Visit 1/Week 1 reactive n=17,4,20 | 7 | 3 | 12
  Visit 1/Week 1 not reactive n=17,4,20 | 8 | 1 | 8
  Visit 1/Week 1 missing value n=17,4,20 | 2 | 0 | 0
  Visit 2/Month 1 reactive n=16,4,20: number analyzed (Participants) | 16 | 4 | 20
  Visit 2/Month 1 reactive n=16,4,20 | 0 | 1 | 14
  Visit 2/Month 1 not reactive n=16,4,20: number analyzed (Participants) | 16 | 4 | 20
  Visit 2/Month 1 not reactive n=16,4,20 | 16 | 3 | 6
  Visit 2/Month 1 missing value n=16,4,20: number analyzed (Participants) | 16 | 4 | 20
  Visit 2/Month 1 missing value n=16,4,20 | 0 | 0 | 0
  Visit 3/Month 6 reactive n=17,4,20 | 4 | 1 | 14
  Visit 3/Month 6 not reactive n=17,4,20 | 11 | 3 | 5
  Visit 3/Month 6 missing value n=17,4,20 | 2 | 0 | 1
  Visit 1 Month after booster reactive n=16,4,18: number analyzed (Participants) | 16 | 4 | 18
  Visit 1 Month after booster reactive n=16,4,18 | 4 | 2 | 15
  Visit 1 Month after booster not reactive n=16,4,18: number analyzed (Participants) | 16 | 4 | 18
  Visit 1 Month after booster not reactive n=16,4,18 | 10 | 2 | 3
  Visit 1 Month after booster missing value n=16,4,18: number analyzed (Participants) | 16 | 4 | 18
  Visit 1 Month after booster missing value n=16,4,18 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from screening visit for a maximum of 69 weeks.
Description: The signing of the Informed Consent was considered the start of treatment for this trial because participants entered the trial on treatment as part of their clinical routine.
Groups:
- Siponimod Continuous: Continuous treatment with siponimod (oral, daily, dose depending on CYP2C9 genotype: 2mg or 1 mg) during SARS-CoV-2 mRNA vaccination
- Siponimod Interrupted: Siponimod (oral, daily, dose depending on CYP2C9 genotype: 2mg or 1 mg) with treatment interruption (for approx. 2-3 months) for the purpose of a SARS-CoV-2 mRNA vaccination
Arm/Group | Siponimod Continuous | Siponimod Interrupted | DMT or No MS Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/4 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/4 | 1/20
Other Adverse Events (participants affected / at risk) | 10/17 | 3/4 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siponimod Continuous (N=17) | Siponimod Interrupted (N=4) | DMT or No MS Treatment (N=20)
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siponimod Continuous (N=17) | Siponimod Interrupted (N=4) | DMT or No MS Treatment (N=20)
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 2
Influenza like illness (General disorders) | 0 | 1 | 2
Injection site erythema (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 3 | 0 | 2
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 4 | 0 | 5
Herpes zoster reactivation (Infections and infestations) | 0 | 0 | 1
Injection site pustule (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1
Body temperature increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Band sensation (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 2 | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04792567/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04792567/SAP_001.pdf